CLINICAL TRIAL: NCT07031752
Title: Impact of Plant-Based Meat Analogues Consumption on Human Health
Brief Title: Plant-Based Meat Analogues and Human Health
Acronym: VegAnimal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government)
Responsible Party: Principal Investigator, MARIO ESTEVEZ, Full Proffesor, Universidad de Extremadura
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 117/2021; MCIN/AEI/10.13039/501100011033 (Other Grant/Funding Number: Spanish Ministry of Science and Innovation)
Record Dates: First submitted 2025-06-04; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Satiation, Satiety; Insulin; Glucose; Leptin Levels; Ghrelin; GLP-1 Concentration; Caloric Intake
Keywords: seitan; beef; satiation; leptin; ghrelin; GLP-1; insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Stage (Experimental): In the first stage, participants were randomly allocated to eat whether vegan meat (VM) or genuine meat (GM) along with water (100 cL).
  Interventions: Other: Postprandial Vegan Meat; Other: Postprandial Meat
- Second Stage (Experimental): The second stage, conducted after a minimum washout period of two weeks following the first stage, was conducted following the same procedure as described for the first stage. Yet, participants shifted positions in relation to the first meal.
  Interventions: Other: Postprandial Vegan Meat; Other: Postprandial Meat

INTERVENTIONS:
Other: Postprandial Vegan Meat — Postprandial responses to one single intake of vegan meat (VM) under fasting conditions.
Other: Postprandial Meat — Postprandial responses to one single intake of genuine meat (GM) under fasting conditions,

SUMMARY:
The goal of this intervention trial is to compare the satiation effects induced by a single intake of vegan meat (VM) and genuine meat (GM) in twenty-five healthy participants, aged 25 to 50 years, from both genders. Participants were randomly allocated to consume either VM or GM along with water during a first sage. In a second stage, conducted following the same procedures as the first after a washout period, participants shifted received the alternative meal (they shifted positions regarding first stage). Blood samples were collected under fasting conditions and at 15, 30, 60 and 120 minutes after meal intake to assess the concentration of glucose, cytokines, leptin, ghrelin, glucagon-like peptide-1 (GLP-1), cholecystokinin (CCK) and insulin. Additionally, urine and feces were collected under fasting conditions at the end of each session.

DETAILED DESCRIPTION:
The study was designed as a postprandial, randomized and crossover intervention trial aimed at comparing the satiation induced by a single intake of grilled vegan "meat" and grilled beef loin at isocaloric and isoprotein conditions. Twenty-five healthy participants (25-50 years old) from both genders (15 females and 10 males) were recruited for the trial and randomly included in a two-stage crossover study. Previously, participants expressed their willingness to participate by signing an informed consent.

In the first stage, participants (fasted during the last 12 hours, without having had a late or heavy dinner, and without engaging in intense physical activity the previous afternoon or evening) were randomly allocated to eat whether vegan meat (VM) or genuine meat (GM) along with water (100 cL). Under fasting conditions, blood samples were collected via venous cannula by clinical nurse collaborators, and the fluids were subsequently treated with a protease inhibitor cocktail by experienced laboratory technicians. Consumption of whether VM or GM was carried out in individual sensory booths at room temperature (22ºC). At fixed postprandial times (i.e., 15, 30, 60 and 120 minutes) blood was collected in dipotassium ethylenediaminetetraacetic acid (K2EDTA) Vacutainer® tubes and treated for the analysis of glucose, cytokines, leptin, ghrelin, GLP-1, CCK and insulin concentrations. During the postprandial period, participants were instructed to remain seated and engage in mild intellectual activity, such as reading a book or working on the computer. Any activity that would interfere with the digestion process or influence the postprandial response to the foods under study was discouraged. Participants were specifically asked not to move around, play games or watch movies. After 120 minutes postprandial time, and in order to assess compensatory caloric intake after the first meal, participants were offered to eat spaghetti Bolognese ad libitum with 100 cL of water until they were fully and comfortably satiated. Caloric intake was recorded by calculating the amount of food had during this ad libitum meal.

The second stage, conducted after a minimum washout period of two weeks following the first stage, was conducted following the same procedure as described for the first stage. Yet, participants shifted positions in relation to the first meal. Researchers and technicians involved in the analysis of samples were blinded to the origin of the samples and the identity of the participants. This information was guarded by an individual unconnected to the study until the completion of the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18-25 kg/m2.
* No clinical signs of metabolic disease (HbA1c < 5.7%).
* Normotensive (<95th centile for height, sex and age).
* Lipid profiles and liver enzymes (aspartate transaminase (AST) and alanine transaminase (ALT)) within physiological range.
* No active medical treatments and no adverse reaction to gluten.

Exclusion Criteria:

* Smoking.
* Drinking alcohol.
* Food allergies.
* Dietary restrictions.
* Not complying with any of the aforementioned requirements

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Plasma glucose levels at predefined postprandial times | At fixed postprandial times after the start of interventions (i.e., 15, 30, 60 and 120 minutes)
  Biochemical profiling of blood samples were carried out in order to analyse glucose concentration at fixed postprandial times
Plasma insulin levels at predefined postprandial times | At fixed postprandial times after the start of interventions (i.e., 15, 30, 60 and 120 minutes)
  Biochemical profiling of blood samples were carried out in order to analyse insulin concentrations at fixed postprandial times
Circulating leptin levels in plasma at fixed postprandial times | At fixed times after the start of interventions (i.e., 15, 30, 60 and 120 minutes)
  Plasma leptin concentration were measured at predefined times after de start of interventions using an enzyme-linked immunosorbent assay (ELISA)-based multiplex assay.
Circulating ghrelin levels in plasma at fixed postprandial times | At fixed times after the start of interventions (i.e., 15, 30, 60 and 120 minutes)
  Plasma ghrelin concentration were measured at predefined times after de start of interventions using an enzyme-linked immunosorbent assay (ELISA)-based multiplex assay.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Extremadura, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT07031752/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT07031752/SAP_001.pdf
  • Informed Consent Form (2022-02-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT07031752/ICF_002.pdf